CLINICAL TRIAL: NCT02080260
Title: A Pilot Study Testing Single-Agent Regorafenib in Advanced Previously-Treated Adenocarcinoma of the Pancreas
Brief Title: A Study of Regorafenib in Advanced Pancreatic Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-GI-PAN-REG-001
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Oral Regorafenib
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — Single agent drug therapy with regorafenib
  Other Names: Stivarga

SUMMARY:
This study tests regorafenib as a single agent in the treatment of metastatic pancreatic cancer patients who have progressed after prior chemotherapy with gemcitabine. The prognosis for these patients is particularly grim, no other standard treatment options exist, and novel approaches are desperately needed.

DETAILED DESCRIPTION:
This is a single arm, single stage Phase II study designed to evaluate progression free survival (PFS) in patients with metastatic pancreatic cancer who have failed at least one prior line of therapy and treatment with gemcitabine. This study is open at the Levine Cancer Institute (LCI). A total of 32 patients will be enrolled over a two years. Following informed consent and eligibility check, all patients will start oral regorafenib therapy (120 mg daily for 3 weeks on / 1 week off; 28 day cycle) with a built-in dose escalation to 160mg after the first cycle as tolerated, and will continue therapy until progression or patient withdrawal. Patients will undergo radiological staging after the first two cycles of regorafenib therapy. Patients with progressive disease will be removed from the study. Patients who have at least stable disease will continue regorafenib therapy, at the Investigator's discretion, and will be radiologically restaged bimonthly.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the exocrine pancreas with metastatic disease.
* The site of the primary tumor confirmed to have been within the pancreas.
* Progression on at least one prior line of chemotherapy for locally-advanced or metastatic pancreatic cancer.
* Progression while on treatment with a gemcitabine regimen for advanced pancreatic cancer, or within 12 months of treatment with gemcitabine as part of adjuvant therapy.
* Measurable disease on axial imaging.
* Age greater than or equal to 18 years.
* Life expectancy of at least 8 weeks.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2. Enrollment of patients with PS = 2 will be capped at 7 patients.
* Subjects must be able to understand and be willing to sign the written informed consent form.
* Acute toxic effects except alopecia of any prior treatment must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 Grade 1 or less.
* Adequate bone marrow, renal, and liver function.
* Warfarin or heparin will be allowed provided that there is no prior evidence of underlying coagulation abnormality.
* Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Patients (men and women) of childbearing potential must agree to use adequate contraception
* Patient must be able to swallow and retain oral medication.

Exclusion Criteria:

* Previous assignment to treatment during this study.
* Uncontrolled hypertension.
* Active clinically significant cardiac disease.
* Cerebrovascular arterial event within 6 months.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any bleeding event greater than or equal to NCI CTCAE Grade 3 within 4 weeks.
* New venous thrombotic or embolic events, such as deep vein thrombosis or pulmonary embolism within 3 months.
* Previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Patients surviving a cancer that was curatively treated and without evidence of disease for more than 3 years are allowed.
* Patients with pheochromocytoma.
* Known history of HIV infection or current chronic or active hepatitis B or C, requiring antiviral medication.
* Ongoing infection greater than or equal to Grade 2 NCI-CTCAE v4.0.
* Symptomatic metastatic brain or meningeal tumors.
* Presence of a non-healing wound, non-healing ulcer, or bone fracture.
* Renal failure requiring dialysis.
* Dehydration Grade greater than or equal to 1 NCI-CTCAE v4.0.
* Patients with seizure disorder requiring medication.
* Persistent proteinuria greater than or equal to Grade 3 NCI-CTCAE v4.0.
* Symptomatic interstitial lung disease.
* Pleural effusion or ascites that cause respiratory compromise.
* History of organ allograft except corneal transplant.
* Known or suspected allergy or hypersensitivity to the study drugs.
* Any severe, uncontrolled malabsorption condition.
* Women who are pregnant or breast-feeding.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study.
* Concurrent anti-cancer therapy other than study treatment (regorafenib).
* Prior use of regorafenib.
* Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days.
* Prior radiation therapy or hepatic arterial therapy is permitted if more than 4 weeks have passed since completion and measurable disease outside of the treated area is present, or if progression since treatment has occurred.
* Use of St. John's Wort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Salmon, MD, Principal Investigator — Atrium Health Levine Cancer Institute; Edward Kim, MD, Principal Investigator — Atrium Health Levine Cancer Institute
Locations (12):
- United States (12):
  - Levine Cancer Institute-Albemarle, Albemarle, North Carolina
  - Levine Cancer Institute-South Tryon, Charlotte, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute - Pineville, Charlotte, North Carolina
  - Levine Cancer Institute - Southpark, Charlotte, North Carolina
  - Levine Cancer Institute - Mallard Creek, Charlotte, North Carolina
  - Levine Cancer Institute - University, Charlotte, North Carolina
  - Levine Cancer Institute - Ballantyne, Charlotte, North Carolina
  - Levine Cancer Institute - Concord, Concord, North Carolina
  - Levine Cancer Institute-Monroe, Monroe, North Carolina
  - Levine Cancer Institute - Cleveland, Shelby, North Carolina
  - Low Country Hematology Oncology, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm, Regorafenib: Oral regorafenib in advanced previously treated pancreatic cancer.
  regorafenib: Single agent drug therapy with regorafenib starting at 120mg per day for 3 weeks out 4, with dose adjustments based upon tolerance
Period: Overall Study
Arm/Group | Single Arm, Regorafenib
Started | 20
Completed | 1 (Defined as still alive in follow-up when the study was terminated and the database was locked.)
Not Completed | 19
Not completed — Death | 18
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Subjects who began regorafenib treatment.
Groups:
- Single Arm, Regorafenib: Oral Regorafenib
  regorafenib: Single agent drug therapy with regorafenib
Arm/Group | Single Arm, Regorafenib
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Progression Free and Surviving at 16 Weeks as a Percent of All Enrolled Subjects
Description: 16-week progression free survival was determined for each subject as a binary variable indicating whether or not the subject is alive and progression free at 16 weeks after treatment start, with progression defined radiographically using RECIST v1.1 or clinically based upon investigator assessment.
Time Frame: 16 weeks after enrollment
Population: Efficacy analyses were conducted on the population of subjects who began regorafenib treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm, Regorafenib
Number analyzed (Participants) | 20
Participants | 2
Statistical Analysis 1: Comparison: Single Arm, Regorafenib; The null hypothesis assumes a median PFS of 6 weeks, corresponding to a 16-week PFS rate of approximately 0.15. A single-stage design will be used to test that the 16-week PFS rate is less than or equal to 0.15. If at least 8 of the 32 subjects are alive and progression free at 16 weeks, the null hypothesis will be rejected. Assuming a one-sided alpha = 0.10 significance level, this will provide at least 90% power to reject the null hypothesis, assuming the true 16-week PFS rate is 0.35; Test type: Superiority; p = 0.824, Fisher Exact — This p-value is only based on partial enrollment of the study. The study enrollment was stopped early due to futility; 16-week PFS Rate = 0.10, 95% CI 2-sided [0.012 to 0.317] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Progression Free Survival
Description: PFS is defined as duration of time from enrollment to the study to time of progression or death. Disease progression (PD) can be objectively determined as per RECIST v1.1 (Response Evaluation Criteria in Solid Tumors, where PD is defined as a 20% increase in the sum of the longest diseased of target lesions, or a measurable increase in non-target lesion, or the appearance of new lesions) or progression can be subjective as determined by the investigator. Evidence for subjective progressions must be documented in medical records. For surviving subjects who do not have documented PD, PFS will be censored at last radiologic assessment. For subjects who receive subsequent anti-cancer therapy prior to documented PD, PFS will be censored at last radiologic assessment prior to commencement of subsequent therapy. Subjects who experience a PFS event following an interval equal to two or more scheduled CT assessments will be censored at date of last assessment prior to first missed assessment.
Time Frame: From date of treatment start to date of progression or death, or censored as described above; assessed for approximately 3 years.
Population: Efficacy analyses were conducted on the population of subjects who began regorafenib treatment
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Single Arm, Regorafenib
Number analyzed (Participants) | 20
weeks | 6.1 [2.9 to 7.1]
Statistical Analysis 1: Comparison: Single Arm, Regorafenib; Test type: Other — Estimation only; Median = 6.1, 95% CI 2-sided [2.9 to 7.1] — The Kaplan Meier method was used to estimate the median PFS(in weeks) for the population. The Greenwood method was used to estimate the confidence limits of the median progression free survival

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration from enrollment date to the date of death from any cause. Subjects who are alive or lost to follow-up at the time of the analysis will be censored at the last known date they were alive.
Time Frame: From date of treatment start to date of death, or censored as described above; assessed for approximately 3 years.
Population: Efficacy analyses were conducted on the population of subjects who began regorafenib treatment
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Single Arm, Regorafenib
Number analyzed (Participants) | 20
weeks | 9.4 [8.1 to 17.0]
Statistical Analysis 1: Comparison: Single Arm, Regorafenib; Test type: Other — Estimation only; Median = 9.4, 95% CI 2-sided [8.1 to 17.0] — The Kaplan Meier method was used to estimate the median OS(in weeks) for the population. The Greenwood method was used to estimate the confidence limits of the median progression free survival

4. Secondary Outcome: Overall Response
Description: Overall response will be determined as the best treatment response for each patient as a binary variable indicating whether or not the patient achieved a Complete Response (CR) or Partial Response (PR) as determined by RECIST v1.1 criteria. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1):Complete Response (CR) is the disappearance of all lesions (target and non target); Partial Response (PR) is at least 30% decrease in the sum of the diameters of target lesions from baseline and no new lesions or unequivocal progression in non target lesions from baseline; Stable Disease (SD) is neither sufficient shrinkage in target lesions to qualify for PR (less than 30% decrease) nor sufficient increase in target lesions (versus smallest sum of diameters) to qualify for PD (less than 20% increase), with no new lesions or unequivocal progression in non target lesions from baseline. For the purposes of response determination, confirmatory scan for CR and PR is not required.
Time Frame: From enrollment to best response while on regorafenib; Subjects remained on treatment until disease progression or death or discontinuation from study or at least 28 days after last dose (subjects were on treatment for an average of 6 weeks)
Population: Efficacy analyses were conducted on the population of subjects who began regorafenib treatment. Analysis of overall response rate was conducted on those patients in the efficacy population with measurable disease present at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm, Regorafenib
Number analyzed (Participants) | 20
Participants | 1
Statistical Analysis 1: Comparison: Single Arm, Regorafenib; Test type: Other — Estimation only; Overall Response Rate = 0.050, 95% CI 2-sided [0.001 to 0.249] — Confidence interval estimated using the Clopper Pearson method

5. Secondary Outcome: Disease Control
Description: Disease control will be determined for each patient as a binary variable indicating whether or not the patient achieved a best overall best response of CR, PR, or stable disease as determined by RECIST v1.1 criteria. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.1): Complete Response (CR) is the disappearance of all lesions (target and non target); Partial Response (PR) is at least 30% decrease in the sum of the diameters of target lesions from baseline and no new lesions or unequivocal progression in non target lesions from baseline; Stable Disease (SD) is neither sufficient shrinkage in target lesions to qualify for PR (less than 30% decrease) nor sufficient increase in target lesions (versus smallest sum of diameters) to qualify for PD (less than 20% increase), with no new lesions or unequivocal progression in non target lesions from baseline.
Time Frame: as for outcome 4
Population: Efficacy analyses were conducted on the population of subjects who began regorafenib treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm, Regorafenib
Number analyzed (Participants) | 20
Participants | 6
Statistical Analysis 1: Comparison: Single Arm, Regorafenib; Test type: Other — Estimation only; Disease Control Rate = 0.300, 95% CI 2-sided [0.119 to 0.543] — Confidence interval estimated using the Clopper Pearson method

ADVERSE EVENTS:
Time Frame: Baseline, during treatment, and 30 days after last dose.
Arm/Group | Single Arm, Regorafenib
All-Cause Mortality (participants affected / at risk) | 18/20
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm, Regorafenib (N=20)
Abdominal pain (Gastrointestinal disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Death NOS (General disorders) | 3
Blood bilirubin increased (Investigations) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Duodenal obstruction (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 — Peritonitis
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other (Infections and infestations) | 2 — bacterial infection, infection & bacteremia
Nausea (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Stroke (Nervous system disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vomiting (Gastrointestinal disorders) | 2
Lung infection (Infections and infestations) | 1
Non-cardiac chest pain (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm, Regorafenib (N=20)
Anemia (Blood and lymphatic system disorders) | 8
Leukocytosis (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
Eye pain (Eye disorders) | 1
Floaters (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Chills (General disorders) | 2
Fatigue (General disorders) | 12
Fever (General disorders) | 5
Pain (General disorders) | 5
Edema limbs (General disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Device related infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 9
Creatinine increased (Investigations) | 3
Investigations - Other (Investigations) | 1 — Elevated blood ammonia level
Lymphocyte count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 6
Weight loss (Investigations) | 8
White blood cell decreased (Investigations) | 3
Hemoglobin increased (Investigations) | 1
Urine output decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 6
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Urinary retention (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Shingles
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT02080260/Prot_SAP_000.pdf